CLINICAL TRIAL: NCT01793935
Title: Sensoril® (Ashwagandha), an Immunomodulator and Anti-inflammatory Agent for Schizophrenia: A Parallel Group, Randomized Double Blind, and Placebo Controlled Study
Brief Title: Withania Somnifera: an Immunomodulator and Anti-inflammatory Agent for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: K.N. Roy Chengappa (Other)
Responsible Party: Sponsor-Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMRI #: 12T-001
Record Dates: First submitted 2013-02-12; First posted 2013-02-18 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Sensoril; Withania Somnifera extract; Total/ Positive / Negative Symptoms; Stress; Inflammation; Immunomodulation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation | interventions — Ashwagandha; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensoril® (Experimental): Sensoril® is a proprietary extract of Withania Somnifera
  Interventions: Drug: Sensoril®
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sensoril® — Sensoril® is a proprietary extract of Withania Somnifera. Each Sensoril® capsules will contain 250 mg of standardized extract of Withania Somnifera
  Other Names: Ashwagandha
  Arms: Sensoril®
Drug: Placebo — Each Placebo capsule comprises inert ingredients; microcrystalline cellulose NF 102, croscarmellose Sodium NF, silicon Dioxide, Fumed NF (Cab-0-sil), magnesium sterate, NF matched in appearance and fill weight to Sensoril® capsules. Moreover, based on past experience, we will expose the placebo capsules to covered sachets containing Sensoril, so that the smell permeates the placebo capsules which then smell like the Sensoril capsules.
  Other Names: "Sugar Pill"
  Arms: Placebo

SUMMARY:
Withania somnifera (WSE; Ashwagandha in Ayurveda) extracts have been used as an adaptogen or to build resistance to stress or diseases in indigenous medical systems in India for centuries. Modern scientific data for WSE indicate several bioactive molecules (withanolides, withanosides, indosides, withaferin-A, others) with significant immunomodulatory, anti-inflammatory and stress reducing properties.

This study will examine whether a standardized extract of Withania Somnifera (WSE; Sensoril®) will improve total, positive, negative symptoms, and stress in patients with schizophrenia. The study will examine whether WSE reduces PANSS positive and negative symptoms and stress scores in subjects, and whether these improvements are mediated by changes in inflammatory immune indices. An additional aim will determine if patients receiving WSE will have fewer adjustments to their psychotropic medications that those assigned to placebo. The study will examine whether WSE will re-balance Th1/Th2 ratios (cytokine measures) and mediate a reduction of elevated hs-CRP levels. It is hypothesized that those subjects whose Th1/Th2 ratios normalize will likely have a greater magnitude of clinical improvement versus those subjects whose immune ratios remain unbalanced.

The proposal is a 12-week, double-blind, placebo-controlled RCT of WSE added to antipsychotic medications in approximately 60 or more patients with schizophrenia with an exacerbation of symptoms. If efficacy is affirmed, this low cost extract could be studied further, and used quite readily across low, middle and high income countries.

DETAILED DESCRIPTION:
The primary aim is to determine whether a standardized extract of Withania somnifera will reduce psychopathology scores (PANSS total) and stress scores(PSS total) in persons with schizophrenia?

The study will also determine whether WSE reduces measures of positive and negative and general symptoms of schizophrenia (PANSS subscale scores)?

Another primary aim will be to determine if changes in antipsychotic and/or other psychotropic medications (lithium, anticonvulsants, antidepressants, anxiolytic agents or hypnotics) (examples: dosage escalation or reductions or switch or stoppage) will favor the group receiving the standardized Withania somnifera extract versus those receiving placebo. Even though we expect changes in antipsychotic medications to occur when patients experience an exacerbation of psychotic symptoms (or other psychiatric symptoms), we hypothesize that those receiving the standardized Withania somnifera extract will experience fewer medication adjustments then those assigned to placebo.

A secondary aim is to determine whether WSE will rebalance TH1/TH2 ratios (cytokine measures) and mediate a reduction of elevated hs-CRP levels? The study will assess whether those subjects whose TH1/TH2 ratios normalize have a greater magnitude of clinical improvement vs. those subjects whose immune ratios remain unbalanced. Similarly, the study will assess whether reduction of hsCRP levels correlate with improvements in PANSS total and subscale scores or the PSS total scores.

Eighty or more patients with DSM IV TR (or if instituted by the study initiation: DSM V) schizophrenia or schizoaffective disorder will be screened and 60 or more eligible patients will be enrolled in a 12 week placebo controlled double blind study. Subjects who have experienced an exacerbation of positive symptoms (delusions, hallucinations, etc). Subjects receiving medications that affect the immune-inflammatory system will be excluded and those receiving antibiotics, antiviral or anti-parasitic medications will be excluded.

Base line laboratory and EKG examination will be carried out to establish eligibility for study participation. In addition specific laboratory analyses of immune markers namely interleukin-2, interferon gamma, interleukin-4, interleukin 6 and high sensitivity C-Reactive Protein will be carried out.

Sixty or more patients will be randomly assigned to receive either WSE or matching placebo starting with 1 capsule of 250 mg strength twice a day (total daily dose = 500 mg) for the first week which will be increased to 2 capsules of 250 mg twice daily (total daily dose = 1000 mg) for a total treatment period of 12 weeks. An assessment of psychopathology (PANSS) and stress will be carried out at each scheduled visit. Assessments of safety including vital signs and treatment emergent adverse events will also be carried out at each visit. Immune-inflammatory markers will be re-assessed at the final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females (≥ 18 years, to 75 years)
2. DSM IV TR diagnosis of schizophrenia or schizoaffective disorder (If officially instituted by study initiation: DSM V diagnoses will be used).
3. Ability to provide informed written consent
4. PANSS total score ≥ 60, positive symptom cluster, (delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility and unusual thought content with at least 2 items scoring ≥ 4, or one of these items scoring ≥ 5, on a scale ranging from 1 = absent to 7 = extreme
5. Current symptom exacerbation ≥ 2 weeks, but ≤ 1 year
6. Receiving anti-psychotic medications for ≥ 4 weeks
7. For women of child bearing age, a negative pregnancy test at screening.

Exclusion Criteria:

1. Testing positive for illicit substances (marijuana or alcohol use will be assessed on a case by case basis, caffeine and nicotine are excepted)
2. Receiving pharmacological treatment for addictions (naltrexone, suboxone, acamprosate, others) will be reviewed on a case by case basis
3. Seriously unstable medical illnesses
4. Pregnant or breast feeding women
5. Known allergy or history of serious adverse event with WSE
6. Subjects who may require imminent hospitalization (examples: suicidal or aggressive behavior)
7. Currently receiving antibiotics, anti-viral, or anti-parasitic medications
8. Currently receiving immunosuppressive medications (e.g. corticosteroids, chemotherapy or transplantation or HIV/AIDs associated drugs).
9. Currently receiving NSAIDs or Aspirin (>81 mg/day) on a daily basis or PRN use > 2x/week (in the last 4 weeks).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KN Roy Chengappa, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Chengappa KNR, Brar JS, Gannon JM, Schlicht PJ. Adjunctive Use of a Standardized Extract of Withania somnifera (Ashwagandha) to Treat Symptom Exacerbation in Schizophrenia: A Randomized, Double-Blind, Placebo-Controlled Study. J Clin Psychiatry. 2018 Jul 10;79(5):17m11826. doi: 10.4088/JCP.17m11826. PMID 29995356

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensoril® | Placebo
Started | 34 | 34
Completed | 28 | 31
Not Completed | 6 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Patient did not take study medication | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 34 subjects were randomized in each group but 1 subject in each group never came to pick up study medication and therefore are not included in the Overall number of participants analyzed in each outcome measure. They did not contribute any data to the intention to treat group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensoril® | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.18 (12.90) | 47.38 (11.37) | 46.28 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 21 | 14 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 14 | 36
  White | 12 | 20 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68
Diagnosis Schizophrenia or Schizoaffective [Count of Participants; unit: Participants]
  Diagnosis Schizophrenia | 21 | 18 | 39
  Diagnosis Schizoaffective | 13 | 16 | 29
Number of lifetime psychiatric hospitalizations [Mean (Standard Deviation); unit: psychiatric hospitalizations] | 7.71 (6.45) | 7.76 (6.90) | 7.74 (6.63)
Age at onset of 1st episode [Mean (Standard Deviation); unit: years] | 24.32 (10.89) | 24.00 (7.67) | 24.16 (9.35)
Current Smokers [Count of Participants; unit: Participants] | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The Positive and Negative Syndrome Scale (PANSS) measures symptom severity in patients with psychotic illnesses. It yields a total score as well as subscores for Positive symptoms, Negative symptoms and General symptoms.
  PANSS Positive subscale consists of 7 Items - (minimum score = 7, maximum score = 49) - Higher values represent a worse outcome.
  PANSS Negative subscale consists of 7 Items - (minimum score = 7, maximum score = 49) - Higher values represent a worse outcome.
  General Psychopathology subscale consists of 16 items - (minimum score = 16, maximum score = 112) - Higher values represent a worse outcome.
  PANSS Total Score - The 3 subscales scores are summed to compute a PANSS Total score. The minimum PANSS total score = 30, maximum = 210 - Higher values represent a worse outcome
Time Frame: Baseline and 12 Weeks
Population: 34 subjects were randomized to each treatment group, but 1 subject in each group did not return to pick up study medication and therefore were not included in the Intention-to-Treat (ITT) sample for analysis of outcomes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale
  PANSS Positive Baseline | 19.58 (3.34) | 19.97 (2.57)
  PANSS Positive at 12 weeks | 14.39 (3.94) | 15.33 (4.75)
  PANSS Negative Baselin | 16.52 (4.52) | 17.27 (5.25)
  PANSS Negative at 12 weeks | 12.97 (4.46) | 15.88 (5.75)
  PANSS General Baseline | 33.79 (5.04) | 33.24 (5.27)
  PANSS General at 12 weeks | 26.55 (4.99) | 30.27 (7.45)
  PANSS Total at Baseline | 69.88 (8.00) | 69.48 (8.45)
  PANSS total at 12 weeks | 53.91 (11.40) | 61.48 (14.89)

2. Secondary Outcome: Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS) was developed to measure the degree to which situations in one's life are appraised as stressful.
  Perceived Stress Scale Scoring Each item is rated on a 5-point scale ranging from never (0) to very often (4). Positively worded items are reverse scored, and the ratings are summed, with higher scores indicating more perceived stress.
  PSS-10 scores are obtained by reversing the scores on the four positive items:
  For example, 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4, 5, 7, and 8 are the positively stated items. Total score can range from 0 to 40. Scores around 13 are considered average. Scores of 20 or higher are considered high stress,
Time Frame: Baseline and 12 weeks or end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale
  PSS score at Baseline | 22.48 (7.27) | 20.55 (6.68)
  PSS score at 12 weeks | 14.67 (5.87) | 18.09 (6.64)

3. Secondary Outcome: Clinical Global Impression Scale (CGI-S) - Severity
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Possible ratings are: 0 = not assessed, 1 = Normal, not at all ill, 2 = Borderline mentally ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Among the most extremely ill patients - The higher the score the worse outcome
Time Frame: Baseline and 12 weeks or end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale
  CGI Severity score at baseline | 4.06 (0.24) | 4.09 (0.38)
  CGI Severity score at 12 weeks | 3.88 (0.49) | 3.97 (0.47)

4. Secondary Outcome: Number of Participants With a Score of 1, 2, or 3 on the Clinical Global Impression Improvement Scale
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: Possible ratings are: 1= Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5= Minimally worse, 6= Much worse, 7=Very much worse.
  The higher the score the worse outcome
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
Participants | 12 | 8

5. Secondary Outcome: Immune Marker IL-2
Description: Changes in immune marker IL-2 will be assessed in response to study medication.
Time Frame: Baseline and 12 weeks or end of study
Population: IL-2 levels undetectable.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
pg/mL | NA (NA) — data cannot be summarized- IL-2 levels undetectable | NA (NA) — data cannot be summarized- IL-2 levels undetectable

6. Secondary Outcome: Immune Marker IL-4
Description: Changes in immune marker IL-4 will be assessed in response to study medication.
Time Frame: Baseline and12 weeks or end of study
Population: Data cannot be summarized- IL-4 levels undetectable
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
pg/mL | NA (NA) — data cannot be summarized- IL-4 levels undetectable | NA (NA) — data cannot be summarized- IL-4 levels undetectable

7. Secondary Outcome: Immune Marker IL-6
Description: Changes in immune marker IL-6 will be assessed in response to study medication.
Time Frame: Changes from Baseline in Immune markers at 12 weeks or end of study
Population: The "number analyzed" differs from the "overall number of participants analyzed" because not all participants had baseline and end of treatment values for IL-6.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
pg/mL
  IL6 level at baseline: number analyzed (Participants) | 30 | 31
  IL6 level at baseline | 3.37 (2.53) | 4.29 (3.34)
  IL 6 level at end of treatment | 3.40 (2.51) | 3.87 (2.57)

8. Secondary Outcome: Immune Marker IFN-Y (Gamma)
Description: Changes in immune marker IFN-Y (gamma) will be assessed in response to study medication.
Time Frame: Baseline and 12 weeks or end of study
Population: data cannot be summarized IFN-Y (gamma) levels undetectable
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
pg/mL | NA (NA) — data cannot be summarized IFN-Y (gamma) levels undetectable | NA (NA) — data cannot be summarized IFN-Y (gamma) levels undetectable

9. Secondary Outcome: Immune Marker Hs-CRP (High Sensitivity C Reactive Protein)
Description: Changes in immune marker hs-CRP (high sensitivity C Reactive Protein) will be assessed in response to study medication.
  hsCRP - mg/L
Time Frame: Baseline and 12 weeks or end of study
Population: The "number analyzed" differs from the "overall number of participants analyzed" because not all participants had baseline and end of treatment values for hs-CRP.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
mg/L
  Pre Rx: number analyzed (Participants) | 30 | 30
  Pre Rx | 5.57 (8.57) | 6.27 (6.90)
  End of Rx | 4.49 (5.09) | 7.82 (8.25)

10. Secondary Outcome: Immune Marker S-100B
Description: Changes in immune marker S-100B will be assessed in response to study medication.
  Elisa
  * Sensitivity 2.7 picogm/ml
  * Range 2.7 to 2000 picogm/ml
Time Frame: Baseline and 12 weeks or end of treatment
Population: The "number analyzed" differs from the "overall number of participants analyzed" because not all participants had baseline and end of treatment values for S-100B.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
pg/mL
  S100B pre Rx: number analyzed (Participants) | 31 | 32
  S100B pre Rx | 39.36 (89.92) | 34.95 (56.12)
  S100B end of Rx | 26.38 (79.44) | 62.49 (173.92)

11. Other Pre Specified Outcome: Vital Signs - Weight
Description: Clinically significant changes in weight will be assessed for "normal" or "abnormal" following randomization to 12 weeks or end of study
Time Frame: Baseline and 12 weeks or end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
lbs
  Body Weight at baseline | 194.61 (49.57) | 191.33 (41.29)
  Body Weight at end of Rx | 197.00 (51.94) | 193.06 (41.33)

12. Other Pre Specified Outcome: Vital Signs - Body Mass Index
Description: Clinically significant changes in BMI will be assessed for "normal" or "abnormal" following randomization to 12 weeks or end of study.
Time Frame: Baseline and 12 weeks or end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
kg/m^2
  BMI at baseline | 30.00 (7.56) | 30.36 (6.35)
  BMI at end of treatment | 30.33 (8.04) | 30.56 (6.24)

13. Other Pre Specified Outcome: Vital Signs - Blood Pressure Systolic and Diastolic
Description: Clinically significant changes in BP will be assessed for "normal" or "abnormal" following randomization to 12 weeks or end of study.
Time Frame: Baseline and 12 weeks or end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
mm/Hg
  Systolic BP at baseline | 124.67 (10.53) | 123.42 (15.32)
  Systolic BP at end of treatment | 123.36 (9.30) | 118.39 (23.19)
  Diastolic BP at baseline | 79.15 (7.95) | 76.52 (11.52)
  Diastolic BP at end of treatment | 79.06 (7.31) | 75.55 (13.21)

14. Other Pre Specified Outcome: Vital Signs - Pulse
Description: Clinically significant changes in Pulse will be assessed for "normal" or "abnormal" following randomization to 12 weeks or end of study.
Time Frame: Baseline and 12 weeks or end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
beats/min
  Pulse at baseline | 76.18 (13.38) | 74.91 (11.75)
  Pulse at end of treatment | 75.42 (14.64) | 76.42 (9.56)

15. Other Pre Specified Outcome: Vital Signs - Temperature
Description: Clinically significant changes in Temperature will be assessed for "normal" or "abnormal" following randomization to 12 weeks or end of study.
Time Frame: Baseline and 12 weeks or end of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees F
Arm/Group | Sensoril® | Placebo
Number analyzed (Participants) | 33 | 33
degrees F
  Temperature at baseline | 97.38 (0.57) | 97.36 (0.72)
  Temperature at end of treatment | 97.37 (0.73) | 97.31 (0.46)

16. Other Pre Specified Outcome: Laboratory Analytes
Description: Changes in laboratory analytes will be classified as "normal" or "abnormal" (example: white blood cell counts)
Time Frame: Change from Baseline in Laboratory Analytes at 12 weeks or end of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were evaluated during the study period (12 weeks)
Description: 34 subjects were randomized to each treatment group, but 1 subject in each group did not return to pick up study medication and therefore were not included in the Intention-to-Treat (ITT) sample for analysis of outcomes
Arm/Group | Sensoril® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 24/33 | 20/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sensoril® (N=33) | Placebo (N=33)
loose stools/diarrhea (Gastrointestinal disorders) | 6 | 5
dry mouth (Gastrointestinal disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 2 | 0
dyspepsia (heartburn) (Gastrointestinal disorders) | 3 | 3
epigastric discomfort (Gastrointestinal disorders) | 3 | 2
anxiety (Psychiatric disorders) | 0 | 2
hyperactive (Psychiatric disorders) | 2 | 0
confusion (Psychiatric disorders) | 0 | 2
worsening of psychiatric symptoms (Psychiatric disorders) | 2 | 1
somnolence (Nervous system disorders) | 7 | 3
headache (Nervous system disorders) | 2 | 4
fatigue/lathargy (General disorders) | 2 | 2
rash (Skin and subcutaneous tissue disorders) | 2 | 0
weight gain (Metabolism and nutrition disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes